CLINICAL TRIAL: NCT02867046
Title: The Incidence of the Intravascular Injection During S1 Transforaminal Epidural Steroid Injection in Two Approaches: Medial vs Lateral in Anteroposterior View
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 4-2016-0442
Record Dates: First submitted 2016-08-07; First posted 2016-08-15 (Estimated); Last update posted 2018-05-18 (Actual); Status verified 2018-05

CONDITIONS: Lumbosacral Radicular Pain
MeSH Terms: interventions — Injections

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- medial approach group (Experimental)
  Interventions: Drug: S1 transforaminal epidural steroid(dexamethasone) injection
- lateral approach group (Active Comparator)
  Interventions: Drug: S1 transforaminal epidural steroid(dexamethasone) injection

INTERVENTIONS:
Drug: S1 transforaminal epidural steroid(dexamethasone) injection — medial approach group (n=85): check intravascular injection while performing S1 transforaminal epidural steroid(dexamethasone) injection in medial side of S1 foramen under fluoroscopy
  lateral approach group (n=85): same as medial approach group except using lateral side of S1 foramen

SUMMARY:
Lumbosacral transforaminal epidural steroid injection (TFESI) is helpful for the treatment of lumbosacral radicular pain, but in case of intravascular injection, infrequently serious complication can be developed. Against this backdrop, if there is any difference of frequency of intravascular injection incidence during S1 (sacrum 1) TFESI between method using medial approach and method using lateral approach in anteroposterior view, the result can be crucial factor in selecting the approach. In addition, appropriate volume of injection will be checked in each approach.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (20-80 years of age) who were scheduled to receive S1 transforaminal epidural steroid injection for lumbosacral radicular pain at pain management clinic

Exclusion Criteria:

1. pregnancy
2. coagulopathy
3. systemic infection
4. any active infection at the injection site
5. history of allergy to contrast media, local anesthetics, corticosteroid
6. patients unable to communicate or patients with cognitive dysfunction

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2016-07-29 (Actual); Primary Completion 2016-11-28 (Actual); Study Completion 2016-11-28 (Actual)

PRIMARY OUTCOMES:
the incidence of intravascular injection in the medial approach group in S1 foramen | 5 seconds after injection of contrast media via block needle.
the incidence of intravascular injection in the lateral approach group in S1 foramen | 5 seconds after injection of contrast media via block needle.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Anesthesia and Pain Research Institute, Yonsei University College of Medicine, Seoul, South Korea